CLINICAL TRIAL: NCT04448314
Title: Study to Evaluate the Usability of PointCheck, a Novel Optical Technology for Screening Non-Invasively Severe Neutropenia
Brief Title: Study to Evaluate the Usability of PointCheck
Status: Completed | Type: Observational
Sponsor: Leuko Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PC001-EU
Record Dates: First submitted 2020-06-10; First posted 2020-06-25 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-03

CONDITIONS: Neoplasms; Chemotherapy-induced Neutropenia
Keywords: Medical Device; Technology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: PointCheck — This is a usability study on PointCheck, a new technology to detect chemotherapy-induced neutropenia

SUMMARY:
This a study about the usability of PointCheck a novel non-invasive technology for monitoring chemotherapy-induced neutropenia. The study will include patients with cancer visiting the outpatient hematology clinic for their standard of care chemotherapy administration. A final sample size of 60 oncologic outpatients will be enrolled and studied with the technology.

The main objective is to evaluate the usability of PointCheck. Secondary outcomes include a preliminary assessment of PointCheck diagnostic accuracy and precision.

For this, study subjects will be tested twice with PointCheck during the same session and the usability in an at-home simulated environment by naïve users will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Study subjects must be able to understand the purpose and risks of the study and to provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations.
2. Male or Female aged 18 years or above
3. Diagnosed with hematological malignancy (e.g., lymphoma, myeloma) or breast cancer.
4. Scheduled active treatment with cytotoxic chemotherapy with an associated high/intermediate risk of neutropenia.
5. Able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria

1. Participants with amputations, congenital malformations or any severe abnormalities of the hands as determined by the investigator.
2. Participants with a history of vasculitis, Raynaud syndrome, scleroderma, mixed connective tissue disease or any other rheumatologic systemic condition that could produce microcirculatory changes in the nailfold.
3. Participants with circulating tumor cells in previous or current lab determinations.
4. Unstable participants or participants with hypotension (systolic blood pressure <90 and diastolic blood pressure < 60mmHg).
5. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
6. Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in participants with malignancies who are scheduled to receive cytotoxic chemotherapy agents with any risk of neutropenia (e.g. antimetabolites, platins, taxanes, topoisomerase inhibitors, Vinca alkaloids, anthracyclines, among others). Participants will be in an ambulatory stable condition as described in the criteria below and according to the investigator's assessment.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
PointCheck's Usability | Up to three-weeks
  To gather data with the ultimate goal of determining the usability of the proposed non-invasive method measured by the the number and % of user errors (globally and per error type) observed in the clinic visits. In addition, the number and % of users successfully completing the test without errors will be measured.
System Usability Scale (0-100 higher scores indicate better usability) | Up to three-weeks
  To confirm the usability of the system using the System Usability Scale

SECONDARY OUTCOMES:
PointCheck's Precision | Up to three-weeks
  To perform an exploratory analysis of the percentage agreement of PointCheck's estimation of WBC from two independent one-minute videos.
PointCheck's Accuracy | Up to three-weeks
  To perform a exploratory analysis of PointCheck's accuracy (e.g., sensitivity, specificity, AUROC) to detect severe neutropenia compared with the gold standard blood analysis method employed by the 12 de Octubre Hospital core laboratory in the range between ≤500 and >500 ANC/µL.
PointCheck's Utility | Up to three-weeks
  To evaluate the % of patients that had to be rescheduled because the sole presence of neutropenia and how many of them were correctly detected with PointCheck.
PointCheck's Safety: total number (%) of AEs and SAEs | Up to three-weeks
  The number (and %) of AEs, SAEs and their relationship with the device use will be the safety endpoint

OTHER OUTCOMES:
Exploratory diagnostic performance for a second cutoff | Up to three-weeks
  The preliminary diagnostic accuracy to detect grade III neutropenia according to CTCAE V5 (<1000 ANC/mm3) 13 measured by the sensitivity and the specificity will be the evaluated with reference to the corresponding laboratory measures acquired.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Martinez López, MD, Principal Investigator — Fundación de Investigación del Hospital 12 de Octubre
Locations (3):
- Spain (3):
  - Hospital Universitari Dexeus. Grupo Quirónsalud, Barcelona
  - Breast Unit. Oncology Department. 12 Octubre Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lamaj G, Pablo-Trinidad A, Butterworth I, Bell N, Benasutti R, Bourquard A, Sanchez-Ferro A, Castro-Gonzalez C, Jimenez-Ubieto A, Baumann T, Rodriguez-Izquierdo A, Pottier E, Shelton A, Martinez-Lopez J, Sloan JM. Usability Evaluation of a Noninvasive Neutropenia Screening Device (PointCheck) for Patients Undergoing Cancer Chemotherapy: Mixed Methods Observational Study. J Med Internet Res. 2022 Aug 9;24(8):e37368. doi: 10.2196/37368. PMID 35943786